CLINICAL TRIAL: NCT02957097
Title: Gabapentin as a Pre-emptive Analgesic in Oral and Maxillofacial Surgical Procedures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Original PI left institution and the PI who took over was not able to initiate the study so it was never started.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff R. Shaefer, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016p001548
Record Dates: First submitted 2016-07-21; First posted 2016-11-07 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Acute Pain; Facial Pain
Keywords: Gabapentin; acute pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Facial Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medication - Gabapentin (Experimental): Participants of this group will be administered either Gabapentin 900 milligram PO 2-3 hours prior to the surgical procedure.
  Interventions: Drug: Gabapentin
- Medication - Placebo (Placebo Comparator): Participants of this group will be administered either Placebo PO 2-3 hours prior to the surgical procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Medication used for management of neuropathic pain conditions
  Other Names: Neurontin; Gralise; Horizant
  Arms: Medication - Gabapentin
Drug: Placebo — Placebo medication. It looks exactly same as the Gabapentin medication in same size, shape, and color.
  Arms: Medication - Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of pre-operative administration of gabapentin 900 mg in management of acute post-operative pain in patients undergoing oral and maxillofacial surgical procedures.

DETAILED DESCRIPTION:
Pain after surgery is a significant acute clinical symptom. It is associated with quality of post-operative recovery, time spent in the hospital, post-discharge care and readmissions, morbidity, psychosocial distress, and cost of care. The management of acute postsurgical pain primarily consists of a multimodal approach consisting of opioids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, and local anesthetics. The associated adverse effects often limit the use of such multimodal pharmacotherapy. Opioids have excellent analgesic properties, however are associated with poor adverse-effects profile. They have been associated with nausea, vomiting, somnolence, and urinary retention. Such adverse-effects may decrease the quality of post-operative recovery, increase patient post-surgical management, and overall cost of care. Moreover, in patients undergoing oral and maxillofacial surgical procedures, such adverse-effects may be further potentiated due to placement of reconstructive plates, screws, and maxillomandibular fixation. In order to improve post-surgical quality of care, researchers have been looking for alternative modalities for the management of acute post-surgical pain. One of such modalities has been use of preemptive analgesic therapy. Preemptive analgesia is defined as a treatment modality that is initiated before a traumatic event, such as, surgical incision or tissue manipulation is introduced. Gabapentin is an antiepileptic drug that has been used in the management of painful neuropathies, such as, diabetic poly-neuropathy, post-herpetic neuralgia, and trigeminal neuropathy. Gabapentin has antiallodynic and antihyperalgesic properties with only a minor effect on normal nociception. It reduces the hyperexcitability of dorsal horn neuron induced by tissue injury, as well as, central sensitization induced after trauma and surgery. Gabapentin has been studied extensively as a preemptive analgesic in various non-craniofacial surgeries. In a systemic review and meta-analysis on the pre-operative administration of gabapentin during various surgical procedures, Tiippana et al reported the opioid-sparing effect during the first 24 h after a single dose of gabapentin 300-1200 mg, administered 1-2 h preoperatively, ranged from 20% to 62%. Authors further concluded that the combined effect of a single dose of gabapentin was a reduction of opioid consumption equivalent to 30 +/- 4 mg of morphine (mean +/- 95% confidence interval) during the first 24 h after surgery. In another meta-regression analysis authors reported that gabapentin reduced opioid related adverse effects, such as nausea, vomiting, and urinary retention (Numbers needed to treat (NNT) 25, 6, and 7, respectively). In a systematic review and meta-analysis, consisting of randomized controlled trials of women who underwent a total abdominal hysterectomy, under general anesthesia, it was concluded that preemptive administration of gabapentin was effective in decreasing postsurgical pain scores, narcotic consumption, and nausea and vomiting episodes. Similar reduction in postsurgical pain scores, narcotic consumption, and adverse effects were seen after other surgical procedures, such as, breast surgery, spinal surgery, orthopedic surgical procedures, and amputation surgery. However, no such data is available for major oral and maxillofacial surgical procedures

Primary and secondary aims are as following:

Primary aims:

1. To determine the difference in the intensity of pain, post-operatively, at 6 hours, 12 hours, 24 hours, and 72 hours between participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.
2. To determine the difference in the total opioid consumption at 24 and 72 hours post-operatively, among participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.
3. To evaluate the difference in the time to first rescue analgesic post-operatively, among participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.
4. To determine the difference in the incidence of adverse effects within first 24 hours and 72 hours post-operatively between participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.

Secondary aims:

1. To determine the difference in the incidence and the intensity of pain at 1 month post-operatively, among participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.
2. To evaluate the differences in post-operative hospital-stay among participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.
3. To evaluate the influence of a history of a chronic pain disorder on:

   1. The association between intensity of pain and pre-emptive use of gabapentin.
   2. The association between opioid consumption and pre-emptive use of gabapentin.
   3. The difference in the time to first rescue analgesic post-operatively, among participants pre-operatively administered gabapentin versus those pre-operatively administered a placebo medication.

Hypothesis:

1. Participants receiving gabapentin 900 mg PO 3h pre-operatively will have significantly less pain at 6 hours, 12 hours, 24 hours, and 72 hours post-operatively compared to those receiving placebo medication.
2. Participants receiving gabapentin 900 mg 3h pre-operatively will have significantly less total opioid consumption at 24 and 72 hours post-operatively than those receiving placebo medication.
3. There will be significantly fewer incidences of adverse events associated with opioid consumption in participants with pre-emptive use of gabapentin medication.
4. The gabapentin group will have significantly longer time to first rescue medication compared to the placebo group.

Study enrollment will be carried out in the department of Oral and Maxillofacial Surgery (OMFS), Massachusetts General Hospital, Boston, Massachusetts. Relevant patients are going to be identified and offered to participate in the study. This will take place during the history and physical examination visit, which is conducted prior to any surgical procedure in the department of OMFS.

This will be a double-blind investigation, randomized, placebo-controlled drug trial. Randomization of treatment group will be carried out by the hospital pharmacy using a computer generated randomization template. Both investigator and participant will be blind to the group allotment.

The investigation is primarily divided into two sections, the medication phase and the surgical phase. In the medication phase of the investigation, treatment group will receive a single dose of Gabapentin 900mg 2-3h before commencement of surgery (initial incision). Placebo group will receive a single dose of placebo medication 2-3h pre-operatively (before commencement of surgery). Both gabapentin and placebo medication will look similar in shape, color, and size. Hospital pharmacy will be recruited to provide the placebo and gabapentin medications. Hospital pharmacy will be responsible for delivering the medication to the participant prior to the surgical procedure.

During the surgical phase of the study, all of the participants will undergo respective oral and maxillofacial surgical procedure, under general anesthesia. The surgical part of this investigation will not, in any way or form, be different than the usual standard of care followed by the department of oral and maxillofacial surgery department, at Massachusetts General Hospital. Peri-operative and post-operative analgesic regimens will also be standardized as per departmental guidelines for the respective surgical procedures.

Data that will be collected consists of following:

Prior to undergoing surgical procedure

1. Age, gender, past medical history, medical illnesses, past surgical history, past hospitalization history, psychosocial history, current medications, allergies.
2. Graded chronic pain scale - 6 months
3. McGill Pain-short questionnaire

After the surgical procedure

1. Surgical characteristics such as, type of surgery, surgeon who performed the surgery, complications during surgery, duration of surgery
2. Pain score on an 11-point likert-type visual analog scale at 6h, 12h, 24h, 72h, 1 month post-surgically.
3. Opioid consumption at 24h and 72h post-operatively
4. Vomiting/Nausea score on an 11-point likert-type visual analog scale at 6h, 12h, 24h, and 72h post-surgically.
5. Opioid-related symptom distress scale at 24h and 72h, post-surgically
6. Duration of hospital stay
7. Analgesic medication regimen after 1 month post-operatively.

All of the data will be collected over 7 data collection points.

Screening phase:

Screening visit. Interested participant will undergo screening and evaluation. Participants will be explained the study and consent will be obtained.

Participants willing to participate will also fill out following questionnaires:

* Graded Chronic Pain Scale 6 months
* McGill pain questionnaire

Surgical phase:

Baseline visit. Participants will be administered either a single tablet of gabapentin 900 mg or a placebo medication, 2-3 hours before undergoing surgical procedure.

Follow-up phase:

Follow-up 1. It will be carried out 6 hours post-surgically. Participant will be asked to rate the level of pain, and intensity of nausea and vomiting on an 11-point likert type 0 to 10 scale, where 0 is indicative of no symptom and 10 is indicative of worst symptom ever. In addition, information from the medical record regarding the characteristics of the surgical procedure (type, surgeon, duration, complications) will be collected.

Follow-up 2, 3, and 4. Follow-up 2, 3, and 4 will be carried out post-operatively, after 12 hours, 24 hours, and 72 hours, respectively. Participant will be asked same questions as in step 3. In addition participants use of analgesic medication and stay in hospital will be recorded. Further more, during follow-up 3 and 4 (24 and 72 hours post-operative, respectively) participants will fill out opioid-related symptom distress scale and data on type, dosage, and quantity of opioid medications consumed will be collected. If participant leaves hospital prior to any of the follow-up visits, they will be contact via telephone.

Follow-up 5. These will be carried out over the phone, at 1 month post-surgically. Following data will be collected:

1. Participants will be asked questions from McGill pain-short questionnaire and opioid-related symptom distress scale.
2. Intensity of nausea and/or vomiting on a 0 to 10 scale, where 0 is indicative of no nausea and/or vomiting and 10 is indicative of worst nausea/vomiting ever.
3. List of analgesic medications.

All types of opioid medications used during the investigation period for management of pain will be converted to morphine sulphate PO equivalent at 0 % cross-reactivity resistance.

BIOSTATISTICAL ANALYSIS

A total of 100 participants are going to be recruited for the present investigation. This number was calculated using either effect size of 25% less consumption of opioid medications, or 25% less pain score at 6h post-operatively, and alpha value of 0.05 and power of 0.95. However, if 100 participants are not recruited by 12 months, recruitment process will be terminated.

A multistep analytic approach will be carried out. In the first step, participants' demographics, and clinical characteristics are going to be compared among participants of the treatment and the placebo group, using t-tests (or non-parametric equivalent) and Chi-squared (or Fisher exact) tests where appropriate. Next, using univariate and multivariate logistic regression analyses are going to be used to determine the efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, of any race, between ages of 18 - 65 years.
2. Participants undergoing unilateral or bilateral Lefort osteotomy, unilateral or bilateral mandibular inverted-L or sagittal split osteotomy with or without genioplasty, temporomandibular joint arthroplasty with or without total joint replacement prosthesis.

Exclusion Criteria:

1. Participants who are pregnant.
2. Participants allergic to gabapentin.
3. Participants with a history of alcohol, or drug abuse.
4. Participants who are unwilling to participate, or are non-compliant to the guidelines of the investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 6 hours postoperatively
  Pain score of participants on a likert type pain scale (0-10), where 0 is indicative of no pain, and 10 indicates worst pain imaginable.
total opioid consumption | 24 hours
  Consumption of opioid medication postoperatively
time to first rescue analgesic | post-operatively (up to 6 hours)
incidence of adverse effects | post-operatively (up to 24 hours)
Intensity of pain | 12 hours postoperatively
  Pain score of participants on a likert type pain scale (0-10), where 0 is indicative of no pain, and 10 indicates worst pain imaginable.
Intensity of pain | 24 hours postoperatively
  Pain score of participants on a likert type pain scale (0-10), where 0 is indicative of no pain, and 10 indicates worst pain imaginable.
Intensity of pain | 72 hours postoperatively.
  Pain score of participants on a likert type pain scale (0-10), where 0 is indicative of no pain, and 10 indicates worst pain imaginable.
total opioid consumption | 72 hours post-operatively
  Consumption of opioid medication postoperatively.

SECONDARY OUTCOMES:
incidence of pain | 1 month
  incidence of pain after 1 month postoperatively
intensity of pain on a numeric rating scale (0-10) | 1 month
  intensity of pain after 1 month post-operative. Pain score of participants on a likert type pain scale (0-10), where 0 is indicative of no pain, and 10 indicates worst pain imaginable.
length of post-operative hospital-stay | postoperatively in terms of days (up to 1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Alayed N, Alghanaim N, Tan X, Tulandi T. Preemptive use of gabapentin in abdominal hysterectomy: a systematic review and meta-analysis. Obstet Gynecol. 2014 Jun;123(6):1221-1229. doi: 10.1097/AOG.0000000000000289. PMID 24807337
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Peri-operative ketamine for acute post-operative pain: a quantitative and qualitative systematic review (Cochrane review). Acta Anaesthesiol Scand. 2005 Nov;49(10):1405-28. doi: 10.1111/j.1399-6576.2005.00814.x. PMID 16223384
- [Background] Dauri M, Faria S, Gatti A, Celidonio L, Carpenedo R, Sabato AF. Gabapentin and pregabalin for the acute post-operative pain management. A systematic-narrative review of the recent clinical evidences. Curr Drug Targets. 2009 Aug;10(8):716-33. doi: 10.2174/138945009788982513. PMID 19702520
- [Background] Marret E, Kurdi O, Zufferey P, Bonnet F. Effects of nonsteroidal antiinflammatory drugs on patient-controlled analgesia morphine side effects: meta-analysis of randomized controlled trials. Anesthesiology. 2005 Jun;102(6):1249-60. doi: 10.1097/00000542-200506000-00027. PMID 15915040
- [Background] Pandey CK, Navkar DV, Giri PJ, Raza M, Behari S, Singh RB, Singh U, Singh PK. Evaluation of the optimal preemptive dose of gabapentin for postoperative pain relief after lumbar diskectomy: a randomized, double-blind, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Apr;17(2):65-8. doi: 10.1097/01.ana.0000151407.62650.51. PMID 15840990
- [Background] Remy C, Marret E, Bonnet F. Effects of acetaminophen on morphine side-effects and consumption after major surgery: meta-analysis of randomized controlled trials. Br J Anaesth. 2005 Apr;94(4):505-13. doi: 10.1093/bja/aei085. Epub 2005 Jan 28. PMID 15681586
- [Background] Gilron I. Is gabapentin a "Broad-spectrum" analgesic? Anesthesiology. 2002 Sep;97(3):537-9. doi: 10.1097/00000542-200209000-00004. No abstract available. PMID 12218517
- [Background] Rose MA, Kam PC. Gabapentin: pharmacology and its use in pain management. Anaesthesia. 2002 May;57(5):451-62. doi: 10.1046/j.0003-2409.2001.02399.x. PMID 11966555
- [Background] Peng PW, Wijeysundera DN, Li CC. Use of gabapentin for perioperative pain control -- a meta-analysis. Pain Res Manag. 2007 Summer;12(2):85-92. doi: 10.1155/2007/840572. PMID 17505569